PRINCIPAL INVESTIGATOR: Hoyoung Maeng, MD

STUDY TITLE: A Pilot Study of Long-Term TARP Vaccination Using a

Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccination in Previously Vaccinated Men on NCI 09-C-

0139

STUDY SITE: NIH Clinical Center

Cohort: Addendum

Consent Version: 10/17/2019

## WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Hoyoung Maeng, MD

240-781-3253

hoyoung.maeng@nih.gov

This addendum provides new information about the study "A Pilot Study of Long Term TARP Vaccination Using a Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccine in Previously Vaccinated Men on NCI 09-C-0139" on which you are enrolled. The information in the consent you signed previously is unchanged.

The NIH Clinical Center Pharmaceutical Development Service (PDS) helps to make the ME TARP DC vaccine used in this study. The PDS was recently closed down by NIH leadership after a vial of contaminated material was discovered on another study just before it was supposed to be given to a research participant. The PDS is undergoing a full review and changes are being made to make sure that processes are in place to prevent anything like this from happening again. The FDA and NIH decided that it might be better and safer to make an exception to the PDS shutdown for some research studies as long as those decisions are made on a case by case or protocol by protocol basis. The ME TARP DC vaccine received one of those exceptions because the parts of the vaccine made by the PDS are just used in the preparation of the vaccine and are never actually given to you, the research participant. Additionally, all of the materials used in making the ME TARP DC vaccine have to pass many tests or they can't be used. Before giving the exception, the FDA and NIH determined that the risk to you from receiving a vaccine that includes the portions made by the PDS, before all of the reviews and changes to the PDS are finished, is extremely low.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Version Date: 10/17/2019

Page 1 of 2

IRB NUMBER: 15C0076 IRB APPROVAL DATE: 12/05/2019

| <u>=</u> | ve read the explanation about this study and have been consent to participate in this study. | given the opportunity |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participant | Date |
| about this study and have been giv<br>to make research decisions on beha | cive (LAR) for an Adult Unable to Consent: I have en the opportunity to discuss it and to ask questions. It all of the adult participant unable to consent and have the the information in the above consent was described to articipate in the study. | am legally authorized e authority to provide |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| | <b>onsent process only:</b> This section is only required if y glish consent form has been approved by the IRB for us | |
| Witness: | | |
| Signature of Witness* | Print Name of Witness | Date |
| *NIH ADMINISTRATIVE SECTION TO BE COMPLETED REGARDING THE USE OF AN INTERPRETER: An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent and served as a witness. The investigator obtaining consent may not also serve as the witness. An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent but did not serve as a witness. The name or ID code of the person providing interpretive support is: | | |
| PATIENT IDENTIFICATION | Consent to Participate in a Clinical Research Stud<br>NIH-2977 (4-17)<br>File in Section 4: Protocol Consent (2)<br>Version Date: 10/17/2019 | ER: 15C0076 |

Page 2 of 2

IRB NUMBER: 15C0076
IRB APPROVAL DATE: 12/05/2019